CLINICAL TRIAL: NCT00476684
Title: The Effect of Radiofrequency-treatment on Patients With Facet-joint Pain in Cervical- and Lumbar-columna
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 023-04REK
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Neck Pain; Low Back Pain
Keywords: radiofrequency
MeSH Terms: conditions — Neck Pain; Low Back Pain | interventions — Pulsed Radiofrequency Treatment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- radiofrequency neurotomy (Experimental): Radiofrequency-neurotomy of the medial branch at 80 degr. C for 70 seconds, after diagnostic blocks
  Interventions: Procedure: radiofrequency treatment
- sham controls (Sham Comparator): Radiofrequency-neurotomy of the medial branch at 37 degr. C needle temperature for 70 seconds, after diagnostic blocks
  Interventions: Procedure: sham neurotomy

INTERVENTIONS:
Procedure: radiofrequency treatment — Radiofrequency-neurotomy of the medial branch at 80 degr. C needle temperature for 70 seconds, after diagnostic blocks
  Arms: radiofrequency neurotomy
Procedure: sham neurotomy — Radiofrequency-neurotomy of the medial branch at 37 degr. C needle temperature for 70 seconds, after diagnostic blocks
  Arms: sham controls

SUMMARY:
There is conflicting evidence on whether radio-frequency neurotomy of the medial branch has a significant effect on pain in patients with chronic unilateral facet joint neck and back pain.

We will evaluate radiofrequency treatment on medial-branch of the ramus dorsalis as an effective pain treatment for patients with chronic pain originated from facet-joints in cervical and lumbar columna.

ELIGIBILITY:
Inclusion Criteria:

* one-sided neck and low back chronic pain
* pain durability of at least 1 year

Exclusion Criteria:

* other somatic or psychiatric disorders
* pregnancy
* stated co-morbidity
* anaesthetics intolerance
* no effect of diagnostic blockades (one or two)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-08 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
reduction in self-reported pain intensity | up to 1 year
  Numerig rating scale 1 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Petter C. Borchgrevink, prof. PhD MD, Principal Investigator — Norwegian University of Science and Technology; Tarjei Rygnestad, Prof. PhD MD, Study Director — Norwegian University of Science and Technology
Locations (1):
- Pain Clinic, University Hospital of Trondheim, Trondheim, Norway